CLINICAL TRIAL: NCT01092195
Title: A Phase I Trial of Safety and Immunogenicity of Gardasil Vaccination Post Stem Cell Transplantation in Patients With and Without Immunosuppression
Brief Title: Gardasil Vaccination in Post Stem Cell Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100083; 10-H-0083
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-07

CONDITIONS: Gardasil Vaccine; Stem Cell Transplant; Immunogenicity
Keywords: Women's Health; Genital Precancer; Stem Cell Donor; Cervical Cytology; Healthy Volunteers; Stem Cell Transplant; Healthy Volunteer; HV
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

ARMS (3):
- Cohort 1 (Active Comparator): Female subjects post stem cell transplant on no systemic immunosuppression. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
  Interventions: Biological: Gardasil
- Cohort 2 (Active Comparator): Female subjects post stem cell transplant with chronic GVHD requiring systemic immunosuppression. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
  Interventions: Biological: Gardasil
- Cohort 3 (Active Comparator): Healthy normal female volunteers. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — 3 separate 0.5 ml intramuscular

SUMMARY:
Background:

* Gardasil , a recently approved vaccine for the sexually transmitted human papillomavirus (HPV), provides immunity to four types of HPV that are associated with genital warts and cervical, vaginal, and vulvar precancer and cancer. The vaccine has been shown to be highly effective in preventing infection with these HPV types and was approved for use by the Food and Drug Administration.
* More research is needed about the vaccine s ability to induce immunity in individuals with suppressed immune systems, such as those who have had other kinds of cancer treatment such as stem cell transplant. Genital warts, precancer, and cancer have been reported as a late complication after stem cell transplant. Researchers are interested in determining whether the HPV vaccine is safe to give and able to induce immunity in female stem cell transplant recipients, their female donors, and healthy female volunteers.

Objectives:

- To assess the safety and immune response of the HPV vaccine in female recipients of stem cell transplants who are either off or on stable doses of immunosuppression.

Eligibility:

* Females between 18 and 50 years of age who have had allogenic stem cell transplants.
* Healthy female volunteers, including stem cell donors, are also eligible for this study.

Design:

* Participants will be screened with a physical examination, blood and urine tests, and saliva samples, and will be asked to complete a sexual quality of life questionnaire.
* Sexually active participants will also have a routine gynecologic evaluation.
* Participants will receive three HPV vaccinations according to the standard vaccination schedule (with the second and third following 2 and 6 months after the first). Participants will record their daily temperature and any reactions to the vaccine on a vaccine report card for 1 week after each vaccination.
* Participants will have clinic visits for further testing 2, 6, 7, and 12 months after receiving the first HPV vaccine.

DETAILED DESCRIPTION:
HPV associated genital dysplasia is a complication following hematopoietic allogeneic stem cell transplantation (HSCT). In a recent study from this institution, one third of female transplant recipients had HPV related genital tract dysplasia. The quadrivalent human papillomavirus virus (HPV) (types 6, 11, 16, 18) vaccine (Gardasil ) is now approved for use in females aged 9-26 for the prevention of cervical cancer and, more recently, vulvar and vaginal cancer. In this study, Gardasil will be used in females age 18 years to 50 at least 90 days post stem cell transplant in two study cohorts to determine its safety and immunogenicity in this population, as a first step to reduce post-transplant HPV-related co-morbidity, genital dysplasia and malignancy. The two study cohorts will both be post transplant; one off of immunosuppression (n=24), and one on immunosuppression (n=24). Gardasil will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months. The primary objectives of this study are to determine the safety and immunogenicity of Gardasil in female allogeneic HSCT recipients. A cohort of healthy subjects will also be vaccinated (n=24) and will serve as a control. Immunogenicity studies characterizing the CD4 and CD8 T- cell response, change in antibody titer and cytokine response from baseline to months seven and twelve will be compared in the three cohorts. Additionally, genital exams will be performed to monitor for HPV. Secondary endpoints will characterize sexual function post-transplant and vulvar/vaginal graft-versus-host disease (GVHD). When available, healthy female stem cell donors corresponding to enrolled vaccine recipients will be enrolled (n=10) as part of the healthy cohort and vaccinated to determine whether there are differences in HPV vaccine immunogenicity in a subset of donors and their respective allogeneic, HSCT female recipients.

As stem cell transplant becomes more applicable to the general population with newer transplant techniques allowing for a larger donor pool and as survival improves, problems associated with long term survivorship such as genital dysplasia, will become more prevalent. Vaccine therapy to prevent or eradicate this disease is needed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Female stem cell transplant recipient at least 90 days post stem cell transplant

OR

Female stem cell transplant recipient at least 90 days post HSCT and on immunosuppression

OR

The matched female stem cell transplant donor for an included stem cell transplant recipient

OR

Healthy female subject

Age greater than or equal to 18 years and less than or equal to 50 years

EXCLUSION CRITERIA:

Vaccine Recipient:

Obvious HPV condyloma or obvious severe dysplasia (greater than or equal to CIN II) warranting treatment

History of severe adverse reaction to any components (yeast, eggs, monosodium glutamate or neomycin) of the quadrivalent HPV vaccine.

Untreated or persistent life-threatening infections not controlled by current treatment

Uncontrolled chronic GVHD i.e. highly active eGVHD requiring immediate intervention

Pregnant or breast feeding or unwilling to be abstinent or practice effective contraception during the study period (note: patients who have been rendered infertile with total body irradiation are eligible)

Enrollment in another vaccine clinical trial during the study period

Enrollment of healthy volunteer in a drug clinical trial during the study period

Inability to comprehend the investigational nature of the study and provide informed consent<TAB>

Prior Gardasil or other HPV vaccination

Persistent or recurrent malignancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Koutsky LA, Galloway DA, Holmes KK. Epidemiology of genital human papillomavirus infection. Epidemiol Rev. 1988;10:122-63. doi: 10.1093/oxfordjournals.epirev.a036020. PMID 2852116
- [Background] Koshiol JE, Laurent SA, Pimenta JM. Rate and predictors of new genital warts claims and genital warts-related healthcare utilization among privately insured patients in the United States. Sex Transm Dis. 2004 Dec;31(12):748-52. doi: 10.1097/01.olq.0000145851.76025.ad. PMID 15608590
- [Derived] Stratton P, Battiwalla M, Tian X, Abdelazim S, Baird K, Barrett AJ, Cantilena CR, Childs RW, DeJesus J, Fitzhugh C, Fowler D, Gea-Banacloche J, Gress RE, Hickstein D, Hsieh M, Ito S, Kemp TJ, Khachikyan I, Merideth MA, Pavletic SZ, Quint W, Schiffman M, Scrivani C, Shanis D, Shenoy AG, Struijk L, Tisdale JF, Wagner S, Williams KM, Yu Q, Wood LV, Pinto LA. Immune Response Following Quadrivalent Human Papillomavirus Vaccination in Women After Hematopoietic Allogeneic Stem Cell Transplant: A Nonrandomized Clinical Trial. JAMA Oncol. 2020 May 1;6(5):696-705. doi: 10.1001/jamaoncol.2019.6722. PMID 32105293
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-H-0083.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant With Immunosuppression: Subjects post stem cell transplant with chronic GVHD requiring systemic immunosuppression. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
- Transplant With no Immunosuppression: Subjects post stem cell transplant on no systemic immunosuppression. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
- Healthy Volunteer: Healthy normal female volunteers. Gardasil® will be administered using the FDA approved regimen of 3 separate 0.5ml intramuscular injections at 0, 2, and 6 months.
Period: Overall Study
Arm/Group | Transplant With Immunosuppression | Transplant With no Immunosuppression | Healthy Volunteer
Started | 23 | 21 | 20
Completed | 23 | 21 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transplant With Immunosuppression | Transplant With no Immunosuppression | Healthy Volunteer | Total
Number analyzed (Participants) | 23 | 21 | 20 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 20 | 64
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 20 | 64
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 12 | 12 | 32
  Black | 11 | 1 | 2 | 14
  Asian | 1 | 5 | 5 | 11
  Hispanic | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Developed Antibody Response to the Vaccine.
Description: The percentage of subjects who developed antibody response to the quadrivalent HPV (qHPV) vaccine (HPV - 6/ - 11/ - 16/ - 18). Anti-HPV-6/11/16/18-specific antibody responses using L1 Virus Like Particle (VLP) ELISA were measured in serum.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant With Immunosuppression | Transplant With no Immunosuppression | Healthy Volunteer
Number analyzed (Participants) | 23 | 21 | 20
Participants | 18 | 20 | 20

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Transplant With Immunosuppression | Transplant With no Immunosuppression | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 23/23 | 18/21 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant With Immunosuppression (N=23) | Transplant With no Immunosuppression (N=21) | Healthy Volunteer (N=20)
Pain (General disorders) | 16 | 14 | 20
Swelling (General disorders) | 6 | 0 | 4
Erythema (General disorders) | 6 | 2 | 5
Pruritus (General disorders) | 3 | 0 | 0
Rash (General disorders) | 1 | 3 | 2
Headache (General disorders) | 1 | 5 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 7 | 4 | 4
Edema (General disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes